CLINICAL TRIAL: NCT06280950
Title: Expanding Liver Transplant Immunosuppression Minimization Via Everolimus (CTOT-43)
Brief Title: Expanding Liver Transplant Immunosuppression Minimization Via Everolimus
Acronym: ELIMINATE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CTOT-43
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Liver Transplant
Keywords: Liver; Transplant; Everolimus
MeSH Terms: interventions — Everolimus; Tacrolimus; Benzocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Interventional Group 1 (Experimental): Participants in this group will slowly reduce their dose of tacrolimus and continue everolimus as their only immunosuppression medication.
  Interventions: Drug: Everolimus; Drug: Tacrolimus (continued reduction)
- Interventional Group 2 (Experimental): Participants in this group will continue to take reduced Tacrolimus and Everolimus IS regimen.
  Interventions: Drug: Tacrolimus (maintain 50% reduction); Drug: Everolimus
- Observational Group (No Intervention): Participants in this group could not tolerate the addition of everolimus. These participants will not be randomized.
  * Participants in this group will stop taking everolimus.
  * Participants in this group will resume taking their tacrolimus +/- mycophenolate compound and prednisone immunosuppression regimen.

INTERVENTIONS:
Drug: Everolimus — * The first step is the addition of everolimus to participants in this group pre-randomization.
  * Participants on a mycophenolate compound will stop taking it within 7 days of initiating everolimus, either by immediate discontinuation or a 7-day taper.
  * Participants taking prednisone will taper off prednisone by 6 months post-transplant.
  * The second step is tacrolimus minimization and withdrawal to everolimus monotherapy in this group after randomization.
  Other Names: Zortress
  Arms: Interventional Group 1
Drug: Tacrolimus (continued reduction) — * Participants randomized in this cohort will have their tacrolimus dose reduced by 50% following randomization.
  * They will maintain this daily dose for 4 weeks/1 month (28-30 days). Tacrolimus withdrawal will occur in intervals of 30 days or 4 weeks.
  * Each subsequent reduction will be based on LFT stability over the prior time interval before the next reduction
  Other Names: FK-506; FR-900506; Prograf; Prograft
  Arms: Interventional Group 1
Drug: Tacrolimus (maintain 50% reduction) — - Participants randomized in this cohort maintain initial reduced dose of Tacrolimus and everolimus for study duration.
  Other Names: FK-506; FR-900506; Prograf; Prograft
  Arms: Interventional Group 2
Drug: Everolimus — * The first step is the addition of everolimus to participants in the interventional group pre-randomization.
  * Participants on a mycophenolate compound will stop taking it within 7 days of initiating everolimus, either by immediate discontinuation or a 7-day taper.
  * Participants taking prednisone will taper off prednisone by 6 months post-transplant.
  * The second step is to continue on the reduced tacrolimus and everolimus regimen.
  Other Names: Zortress
  Arms: Interventional Group 2

SUMMARY:
This is a study to determine the safety, efficacy, and tolerability of taking away the anti-rejection medicine, tacrolimus, in liver transplant recipients in conjunction with everolimus monotherapy to preserve renal function. Two hundred - seventy (270) subjects will be randomized 2:1 into one of two groups between 2-3 months post-transplant. Seventy participants will be placed into an observational group and will remain on their current post-transplant medications. The duration of the study from time of enrollment is 18-20 months.

DETAILED DESCRIPTION:
This study is a multicenter 2:1 randomized nonblinded phase II interventional clinical trial in liver transplant recipients. The primary objective is to determine the safety, efficacy, and tolerability of tacrolimus minimization and eventual withdrawal in conjunction with everolimus monotherapy to preserve renal function. Study subjects will undergo first reduction of tacrolimus with the addition of everolimus. If everolimus is tolerated, subjects will be randomized 2:1 into one of two interventional arms. The first interventional arm will undergo a stepwise reduction of tacrolimus and be on everolimus monotherapy for the remainder of the study. The second interventional arm will remain on the initial reduced tacrolimus dose and everolimus. If subjects prior to randomization are unable to tolerate everolimus, these subjects will be placed in the observational group. These subjects will stop taking everolimus and resume their immunosuppression therapy prior to study enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject and/or legal guardian must be able to understand and provide informed consent
2. Adult (age greater than or equal to 18 years of age at time of informed consent) recipient of first liver transplant alone (de novo)
3. Estimated glomerular filtration rate >=30 ml/min/1.73m^2 at enrollment using the CKD-EPI 2021 equation
4. Treatment with tacrolimus therapy, with or without mycophenolic acid derivatives and/or corticosteroids
5. Female subjects of childbearing potential with negative pregnancy test upon study entry
6. All subjects of reproductive potential agreeing to use contraception for the duration of the study
7. Previous vaccination or documented immunity to varicella, measles, hepatitis B, pneumococcus, influenza, zoster (if >=19 years old), and 2019-nCoV (COVID-19) as outlined in the DAIT Vaccination Guideline

Exclusion Criteria:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol
2. Active unresolved systemic viral, bacterial, fungal, or parasitic infection requiring oral or intravenous anti-infective therapy
3. History of autoimmune liver disease including autoimmune hepatitis, primary sclerosing cholangitis, and/or primary biliary cirrhosis, or other contraindications to drug withdrawal
4. History of non-hepatic autoimmune disease requiring current or future systemic immunosuppressive therapy other than per study protocol
5. History post-transplant of Hepatic Artery Thrombosis or Portal Vein Thrombosis.
6. History of recurrent cirrhosis after liver transplantation.
7. Chronic use of systemic glucocorticoids, biological immunomodulatory therapy, or other immunosuppressive agents other than per study protocol
8. History of hepatitis B or C virus infection with detectable viral PCR at enrollment
9. History of prior organ transplantation (liver or other type)
10. History of >= 2 biopsy-proven acute cellular rejection episodes of any severity, >=1 moderate to severe rejection episode (histologically defined or requiring lymphodepletion therapy), or >= 1 antibody- mediated rejection episode
11. Active treatment with any mTOR-inhibitor agent (everolimus, sirolimus)
12. Contraindication to treatment with everolimus (open wound or wound infection; urine protein: creatinine ratio > 0.5; significant pancytopenia (any of the following: WBC <1.5 K/uL or ANC <1000 cells/uL or actively being treated with GCSF; Hb <8.0; platelet count <50K); serum triglycerides > 1000 mg/dL; other per PI)
13. Abnormal liver function tests on study entry: Total Bilirubin (TB)>1.5 mg/dL and Direct Bilirubin (DB) >1.0 mg/dL, Alkaline Phosphatase (AP) >200 U/L, and Alanine Aminotransaminase (ALT)>60 U/L
14. Pregnant on enrollment or plan to become pregnant during the study period
15. Participation in another clinical trial that would interfere with this study's procedures and intervention:

    1. Use of investigational biologic or drug (within 8 weeks of study enrollment)
    2. Additional blood collection that would exceed research blood draw limits
    3. Any other procedure or intervention, in the investigator's opinion would interfere with this study
16. Received live attenuated vaccine(s) within 2 months of enrollment
17. Current, diagnosed, mental illness or current, diagnosed, or self-reported drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study
18. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Percent change in estimated glomerular filtration rate (eGFR) by CKD-EPI 2021 equation. Between Cohorts INT-1 and INT-2 | From Visit 2 to Visit 9 (12 months post-liver transplant)
Proportion of subjects with treated Biopsy Proven Acute Rejection (tBPAR) per local pathology. Between cohorts INT-1 and INT-2 | From Visit 2 to Visit 9 (12 months post-liver transplant)

SECONDARY OUTCOMES:
Percent change in estimated Glomerular Filtration Rate (eGFR) | From Visit 1 to Visit 11 (20 months post-liver transplant)
Percentage of subjects with treated Biopsy Proven Acute Rejection (tBPAR) | From Visit 1 to Visit 11 (20 months post-liver transplant)
Changes in liver graft function: Total bilirubin | From Visit 1 to Visit 11 (20 months post-liver transplant)
Changes in liver graft function: Direct bilirubin | From Visit 1 to Visit 11 (20 months post-liver transplant)
Changes in liver graft function: Alanine Aminotransaminase (ALT) | From Visit 1 to Visit 11 (20 months post-liver transplant)
Changes in liver graft function: Aspartate Aminotransferase (AST) | From Visit 1 to Visit 11 (20 months post-liver transplant)
Changes in liver graft function: Alkaline Phosphatase | From Visit 1 to Visit 11 (20 months post-liver transplant)
Time to graft failure in liver function defined as relisting for transplantation, re-transplantation itself or death with failed graft | From Visit 1 to Visit 11 (20 months post-liver transplant)
Time to all-cause mortality | From Visit 1 to Visit 11 (20 months post-liver transplant)
Proportion of subjects experiencing a Major Adverse Cardiac Event (MACE) | From Visit 1 to Visit 11 (20 months post-liver transplant)
Proportion of subjects experiencing infection requiring hospitalization | From Visit 1 to Visit 11 (20 months post-liver transplant)
Proportion of subjects experiencing any malignancy | From Visit 1 to Visit 11 (20 months post-liver transplant)
Proportion of subjects developing severe Estimated Glomerular Filtration Rate (eGFR) deterioration >40 percent from baseline using the CKD-EPI 2021 equation | From Visit 1 to Visit 11 (20 months post-liver transplant)
Proportion of subjects developing any major immunosuppressive therapy complications | From Visit 1 to Visit 11 (20 months post-liver transplant)
Proportion of subjects developing new onset peripheral edema | From Visit 1 to Visit 11 (20 months post-liver transplant)
Proportion of subjects developing new onset cytopenia deemed WBC <3.0x10^9 /L, Hb <8.0 g/dL, or platelets <50 x 10^9/L. | From Visit 1 to Visit 11 (20 months post-liver transplant)
Proportion of subjects developing new onset oral/gastrointestinal ulcerations | From Visit 1 to Visit 11 (20 months post-liver transplant)
Proportion of subjects developing new onset gastrointestinal symptoms (nausea, vomiting, abdominal pain, or diarrhea) related to everolimus therapy. | From Visit 1 to Visit 11 (20 months post-liver transplant)
Proportion of subjects developing new onset pneumonitis | From Visit 1 to Visit 11 (20 months post-liver transplant)
Proportion of subjects developing new onset hepatic artery thrombosis | From Visit 1 to Visit 11 (20 months post-liver transplant)
Proportion of subjects developing other adverse events deemed | From Visit 1 to Visit 11 (20 months post-liver transplant)
Proportion of subjects developing any adverse events related to everolimus therapy | From Visit 1 to Visit 11 (20 months post-liver transplant)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Boike, MD, Principal Investigator — Northwestern University Feinberg School of Medicine: Transplantation
Locations (8):
- United States (8):
  - Mayo Clinic Hospital Arizona (Site #: 71144), Phoenix, Arizona
  - University of California, San Francisco (Site #: 71108), San Francisco, California
  - Northwestern University (Site #: 71110), Chicago, Illinois
  - Icahn School of Medicine at Mount Sinai (Site #: 71115), New York, New York
  - Duke University Medical Center (Site #: 71139), Durham, North Carolina
  - University of Pennsylvania (Site #: 71111), Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (Site #: 71170), Pittsburgh, Pennsylvania
  - Baylor Medical Center (Site #: 71153), Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 24 Months after database lock for the trial
Access Criteria: Open Access
URL: http://www.immport.org/home